CLINICAL TRIAL: NCT05888870
Title: The Outcome Comparison of Immune Tolerance Induction Therapy Using SCT800 Combined With Daratumumab or SCT800 Alone in Hemophilia A Adolescents and Adults With High Titer Inhibitor: a Non-randomized Controlled Trial
Brief Title: ITI Using SCT800 Alone or Combining Daratumumab in Hemophilia A Adolescents and Adults With High Titer Inhibitor
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022035
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia A With Inhibitor
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCT800 combined with Daratumumab (Experimental): ITI using low-dose domestic rFVIII (SCT800) (50IU/kg TIW) and treated with Daratumumab 8mg/kg 4-8 times. Other immunosuppressants could be added after 3 months.
  Interventions: Drug: SCT800 and Daratumumab
- SCT800 alone (Active Comparator): ITI using low-dose domestic rFVIII (SCT800) (50IU/kg TIW) alone. Other immunosuppressants could be added after 3 months.
  Interventions: Drug: SCT800

INTERVENTIONS:
Drug: SCT800 and Daratumumab — SCT800 50IU/kg TIW alone or treated with Daratumumab 8mg/kg 4-8 times
  Other Names: Immune tolerance induction combine anti-CD38
  Arms: SCT800 combined with Daratumumab
Drug: SCT800 — SCT800 50IU/kg TIW alone
  Other Names: Immune tolerance induction only
  Arms: SCT800 alone

SUMMARY:
To evaluate the time of response, sustained remission rate, and relapse rate of CD38 monoclonal antibody (Daratumumab) combined with SCT800 (rFVIII) in the treatment of hemophilia A adolescents and adults with high titer inhibitors.

DETAILED DESCRIPTION:
This is a non-randomized controlled trial to compare the outcome of immune tolerance induction therapy usingnon- SCT800 combined with Daratumumab or SCT800 alone in hemophilia A adolescents and adults with high titer inhibitors. Patients will receive Daratumumab combined with SCT800 or SCT800 alone.

ELIGIBILITY:
Inclusion Criteria

1. Moderate or severe hemophilia A;
2. Aged 14-66 years old;
3. Inhibitor positive at 2 consecutive visits;
4. Inhibitor titer > 10 BU at the screening visit.

Exclusion Criteria:

1. The patient has contraindications to drug ingredients or hamster protein allergy;
2. Suffering from other immune diseases or Using immunosuppressant IS to treat another disease(s);
3. Failed systemic ITI treatment in history;
4. Poor patients compliance;
5. The investigator believes that there are any other reasons that make the patient unsuitable to participate in this study.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
success rate of ITI success rate of ITI success rate of ITI success rate of ITI | 12 months
  Inhibitor titre <0.6 BU⁄mL
Success rate and partial success rate of ITI after 3-month treatment | 3 months
  Inhibitor titre <0.6 BU⁄mL

SECONDARY OUTCOMES:
ITI success time | 12 months
  time to successful tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital; Renchi Yang, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
Data can be requested from the corresponding authors from 12 months to 36 months after study completion
Supporting Information: Study Protocol
Time Frame: from 12 months to 36 months after study completion
Access Criteria: From corresponding author